CLINICAL TRIAL: NCT05208710
Title: A First-in-human, Phase I, Single-center, Open-label, Dose-escalation Trial in Healthy Volunteers to Assess Safety, Tolerability, and Immunogenicity of PANHPVAX, a Vaccine Targeting Human Papilloma L2 Antigen Formulated With Cyclic Di-AMP
Brief Title: PANHPVAX, Study of a New HPV Vaccine in Healthy Volunteers
Acronym: PANHPVAX
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other); National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: DKFZ-2019-003; 2021-002584-22 (EudraCT Number)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: HPV
Keywords: HPV Vaccines; Cyclic-di AMP; First in Human
MeSH Terms: interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PANHPVAX 10µg (Experimental): PANHPVAX 10µg plus c-di AMP in escalating doses
  Interventions: Biological: Vaccination with PANHPVAX 10µg
- PANHPVAX 40µg (Experimental): PANHPVAX 40µg plus c-di AMP in escalating doses
  Interventions: Biological: Vaccination with PANHPVAX 40µg
- PANHPVAX 100µg (Experimental): PANHPVAX 100µg plus c-di AMP in escalating doses
  Interventions: Biological: Vaccination with PANHPVAX 100µg

INTERVENTIONS:
Biological: Vaccination with PANHPVAX 10µg — Escalated dosages of c-di AMP (0, 7,5, 15µg) added groupwise to 10µg antigen
  Arms: PANHPVAX 10µg
Biological: Vaccination with PANHPVAX 40µg — Escalated dosages of c-di AMP (0, 7,5, 15µg) added groupwise to 40µg antigen
  Arms: PANHPVAX 40µg
Biological: Vaccination with PANHPVAX 100µg — Escalated dosages of c-di AMP (0, 7,5, 15µg) added groupwise to 100µg antigen
  Arms: PANHPVAX 100µg

SUMMARY:
First-in-human, phase I, single-center, open-label, dose-escalation trial in healthy volunteers. Investigation of safety and tolerability of ascending doses of PANHPVAX, a vaccine against human papilloma L2 antigens formulated with cdA (adjuvant) as compared to the formulation without cdA.

DETAILED DESCRIPTION:
Infections with one of 15 human papillomavirus (HPV) types are considered the main risk factor for the development of certain anogenital cancers. In addition, these HPV types are also suspected to be causatively involved in oropharyngeal cancer. Three commercial vaccines are currently available, which are inducing prophylactic neutralizing antibody responses against the L1 major capsid protein. The vaccines are cocktails of L1 virus-like particles of two to nine different HPV types. L1 is not preserved between serotypes, therefore, the specific immune responses, are limited to the HPV types represented by the vaccine. In contrast, the L2 minor capsid protein harbors a so called major cross-neutralization epitope in its amino terminus, which has a high homology between serotypes. The PANHPVAX vaccine is based on this epitope.

Specifically, a polytope containing the epitope of eight HPV types is inserted into a scaffold of thioredoxin from the archaeon Pyrococcus furiosus. Further, the antigen is multimerized by a heptamerization domain. To increase immunogenicity, the protein is formulated with the di-nucleotide adjuvant cyclic di-adenosine monophosphate (used abbreviations: cyclic di-AMP / c-di-AMP/ cdA), an inducer of cellular STING (Stimulator of Interferon Genes). In preclinical models, PANHPVAX induces neutralizing antibodies against all cancer-causing HPV types as well as the major types causing benign genital warts. Also, neutralizing antibodies are induced against a number of cutaneous HPV that are suspected to play a role in skin carcinogenesis and/or cause morbidity in immunocompromised patients.

The investigators aim to translate the vaccine into clinical use and conduct a first-in-human single-center dose-escalation trial in healthy volunteers with an intramuscular (i.m.) prime and two i.m. booster injections to demonstrate safety, tolerability, and immunogenicity of the PANHPVAX antigen. The vaccine will be administered in escalating doses and with increasing amount of the adjuvant cdA (novel excipient) in the formulation, in each dose cohort starting with a group of volunteers who will receive the vaccine without adjuvant. Individual participants will be treated three times with identical doses at months 1, 3, and 6 and followed up for safety and tolerability. Induction of neutralizing antibody responses will be determined by pseudovirion-based neutralization assay (PBNA), the current gold standard for monitoring HPV prophylactic vaccines.

Volunteers will be vaccinated with PANHPVAX antigen, reconstituted for administration with novel excipient cdA as adjuvant and dilution buffer. Each volunteer is scheduled to receive three identical vaccine doses. The initial (prime) vaccination is followed by two booster vaccinations one and six months thereafter (Figure 1). After each administration, a close follow-up for vaccination reactions will occur for 29 ± 3 d and a long-term safety follow-up will be scheduled about 13 months after the first vaccine dose (= 6 months after the last vaccine dose).

Dose-escalation cohorts are defined by the antigen dose. Within each cohort, three dose groups of volunteers will receive the vaccine with escalating doses of adjuvant (no adjuvant/0 µg, 7.5 µg, and 15 µg cdA) in the formulation, always starting with a group of 3 volunteers who will receive PANHPVAX formulated without adjuvant. This is followed by two consecutive groups of 6 volunteers each receiving the same antigen dose in combination with ascending doses of adjuvant.

After the first administration of each dose combination of antigen and adjuvant ("prime"), safety observation periods will be longer and the first two participants in each dose group will be exposed separately. Thereafter, all further volunteers of a group may be dosed in parallel. In the two subsequent boosting phases, 2 participants per dose group are planned to be exposed first and observation periods between subsequent enrolment will be slightly shorter. New dose cohorts may be opened as soon as the data safety monitoring board (DSMB) assessed the safety data available after the 15th participant of a cohort has received his/her second vaccine administration (= 1st boost) and has been observed for 7 d.The DSMB will evaluate the data and provide its recommendation on continuation.

ELIGIBILITY:
Inclusion Criteria:

1. Written, personally signed and dated informed consent to participate in the trial prior to any trial-related interventions,
2. Understanding, ability, and willingness to fully comply with trial interventions and restrictions,
3. Age 18-45 years (y) inclusive at the time of consent,
4. Males or females of child-bearing potential who are willing to use a highly effective method of contraception during the treatment and for 4 weeks after each vaccination with the IMP, or women not of child-bearing potential (WNCBP), or individuals who are convincingly sexually abstinent. Highly effective methods of contraception are described in section 7.6.9,
5. No current desire to have children, and
6. Consent not to be vaccinated with a commercially available HPV vaccine during the trial until the end-of-study visit.

Exclusion Criteria:

1. Clinically significant or relevant abnormalities as assessed by the investigator in the medical history, or findings from physical examination, or laboratory evaluation that may require treatment or make the participant unlikely to fully complete the trial, or any condition that presents undue risk from the IMP or trial interventions,
2. Any acute or chronic illness expected to influence the immune response to vaccination,
3. Immunoglobulin administration in the past 3 months prior to first immunization,
4. Any known history of severe anaphylactic reactions to drugs or vaccinations, or any known history to allergies against the excipients of the investigational medicinal product (IMP),
5. Clinically relevant findings in any of the following investigations at screening (SCR) I. Hemoglobin (Hb) < 12 g/dl (males) or < 11 g/dl (females), II. Estimated Creatinine clearance (eCrCl) < 60 ml/min (Cockcroft-Gault), III. Total bilirubin > upper limit of normal (ULN) x 1.2; In case of suspected Gilbert´s disease: total bilirubin ≤ ULN x 3 is acceptable , IV. Alanine aminotransferase (ALT) > ULN x 1.1, V. Aspartate aminotransferase (AST) > ULN x 1.2,
6. Use of an IMP within 30 d prior to the expected date of receiving the first dose of IMP or active enrolment in another drug or vaccine clinical trial,
7. Use of any medication (prescription medication, non-prescription medication including herbal preparations) with active ingredients (except hormonal contraception, iodine, and thyroid hormones) within a period of less than 5 times the respective elimination half-life (t1/2) with regard to the expected date of the first dose of IMP. This does not apply to topical preparations if no relevant systemic exposure is expected,
8. Known prior vaccination against HPV,
9. Any vaccination within the 28 days (d) prior to the expected Visit 1,
10. A positive human immunodeficiency virus (HIV) or hepatitis C (HCV) antibody screen, or positive result for Hepatitis-B-Surface-Antigen (HBsAg),
11. A positive result in the drug screening test at SCR, and
12. Pregnancy or breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of local and systemic reactions | 3 months
  Frequency and severity of local and systemic reactions (solicited vaccination reactions) of ascending doses of the vaccine after each vaccination until day 29.

CONTACTS AND LOCATIONS:
Overall Officials: Antje Blank, Dr., Principal Investigator — Heidelberg University Hospital, Department of Clinical Pharmacology and Pharmacoepidemiology
Locations (1):
- University Hospital Department of Clinical Pharmacology and Pharmacoepidemiology, Heidelberg, Germany